CLINICAL TRIAL: NCT00174590
Title: Treatment of Major Depressive Disorder With Psychotic Features With Risperidone Monotherapy; Risperidone and Sertraline; or Haloperidol and Sertraline
Brief Title: Treatment of Major Depressive Disorder With Psychotic Features.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIS-USA-248; RIS-USA-248
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Major Depression With Psychotic Features
Keywords: depression
MeSH Terms: conditions — Depression | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to determine the safety and efficacy of risperidone monotherapy in the treatment of psychotic depression. We hypothesize that risperidone is as equally as effective as haloperidol plus sertraline for depression with psychotic features

DETAILED DESCRIPTION:
Risperidone is a novel antipsychotic that is usually not associated with the adverse effects of neuroleptics. In addition, preliminary evidence suggests that it has additional mood stabilizing properties as compared with neuroleptics. We are examining the effect of risperidone alone for the treatment of psychotic depression. After providing written informed consent, subjects with major depression and psychosis will undergo a routine medical and neurological evaluation. If subjects qualify they will undergo a 3 to 7 day washout. Subjects will be randomly assigned under double-blind conditions to risperidone plus placebo; risperidone plus sertraline; or haloperidol (HPDL) plus sertraline in a prospective parallel design for a 6 week trial. Outcome measures include the Hamilton Rating Depression Scale, The Positive and Negative Symptom Scale and the Clinician Administered Ratings Scale for Mania and Simpson Angus Scale. Rating will be conducted on a weekly basis throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be men and women 18 to 70 years of age with major depression and psychosis that is either an initial episode or a recurrent episode (unipolar or bipolar).
* Subjects with an anxiety disorder or an additional mood disorder such as dysthymia are eligible.
* Baseline HDRS score of greater than 21.
* A baseline PANSS score of greater than 4 on at least one of the 5 psychosis items

Exclusion Criteria:

* Pregnant women Women of child-bearing age who refuse a urine pregnancy test or who refuse to use a contraceptive technique when sexually active.
* Persons with other psychotic disorders; a mood disorder due to a general medical condition or substance-induced; a current substance dependence disorder; or a dementing disorder are excluded.
* Persons with serious, unstable medical illnesses.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale

CONTACTS AND LOCATIONS:
Overall Officials: Philip g Janicak, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States